CLINICAL TRIAL: NCT01467453
Title: Clinical Application of Sensimed Triggerfish Sensor (TS) With Wireless Signal Transmission for Continuous Intraocular Pressure Measurement
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Triggerfisch-001
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: Triggerfish — The Triggerfish is a contact lens with an embedded sensor to track changes in intraocular pressure during a period of 24 hours.
  Other Names: Triggerfish, SENSIMED AG, Route de Chavannes 37, 1007 Lausanne, Switzerland

SUMMARY:
The study objective is to investigate the clinical applicability of continuous IOP measurement using TS with radio transmission over 24 hours.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of glaucoma

Exclusion criteria:

* Other opticus neuropathy than glaucoma
* Corneal abnormalities (e.g. scaring)
* Dry eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Study Completion 2012-12

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Christoph Kniestedt, Assistant Prof, MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Switzerland